CLINICAL TRIAL: NCT03957993
Title: Pilot Study: Addressing Home-Based Functional Challenges Via Telehealth-Based Occupational Therapy
Brief Title: OT Intervention Via Telehealth for Children With ASD and ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-5623
Record Dates: First submitted 2019-05-10; First posted 2019-05-21 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the Telehealth arm of the study or the Standard Care arm of the study.
Who Masked: Outcomes Assessor
Masking Description: The therapist who assesses the outcomes is a different therapist than the treating (intervention) therapist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational Therapy via Telehealth (Experimental): Participants in the telehealth-based model will undergo occupational therapy treatment via a telehealth-based video chat platform for the entire episode of care (generally 10-12 weeks in duration). The patient will use the video chat client to connect to his/her occupational therapist, and the therapist will conduct the session over this virtual connection.
  Interventions: Other: Occupational Therapy via Telehealth
- Standard of Care Occupational Therapy (Active Comparator): Participants in the standard of care model will undergo occupational therapy treatment via traditional in- person encounters in an outpatient clinic setting for the entire episode of care (generally 10-12 weeks). These children will receive routine occupational treatment via in-person sessions with an occupational therapist conducted in an outpatient clinic setting.
  Interventions: Other: Standard of Care Occupational Therapy

INTERVENTIONS:
Other: Occupational Therapy via Telehealth — The caregiver will be with the participant in their home environment receiving occupational therapy via Telehealth (video-calling) with the occupational therapist.
  Arms: Occupational Therapy via Telehealth
Other: Standard of Care Occupational Therapy — The caregiver and participant will be in the clinic receiving occupational therapy in-person with the occupational therapist.
  Arms: Standard of Care Occupational Therapy

SUMMARY:
This study aims to measure the impact of a telehealth-based model of occupational therapy (OT) treatment on clinical outcomes for children with autism spectrum disorder (ASD) and/or attention deficit hyperactivity disorder (ADHD). Half of the participants will receive clinic-based, in-person services and half of the participants will receive video-based, Telehealth services.

DETAILED DESCRIPTION:
Children with autism spectrum disorder (ASD) and/or attention deficit hyperactivity disorder (ADHD) often receive occupational therapy (OT), which traditionally takes place in a clinical setting. This setting may present barriers and distractors that make it hard for children to achieve their OT goals. Telehealth-based sessions provide an alternative, allowing the therapist to be virtually present within the home.Once enrolled, children will randomly be assigned to be in one of two groups: (1) Standard, in which children will receive clinic-based services as per standard of care OR (2) Telehealth, in which children will receive in-home services on a video-based platform on a timeline identical to what they would receive if they were in the Standard group. Children in both groups will participate for the duration of the episode of care, estimated to last 10-12 weeks. Assessments will be completed at initial evaluation, discharge, and three months following discharge.

ELIGIBILITY:
Inclusion Criteria:

* Has a Autism Spectrum Disorder and/or Attention Deficit Hyperactivity Disorder
* Has an active occupational therapy referral
* Has occupational therapy goals that are directly related to performance of activities of daily living that might reasonably be affected by the environment (as determined by an evaluating therapist)

Exclusion Criteria:

* Does not have Autism Spectrum Disorder or Attention Deficit Hyperactivity Disorder
* Does not have an active occupational therapy referral
* Does not have occupational therapy goals that are directly related to performance of activities of daily living that might reasonably be affected by the environment (as determined by an evaluating therapist)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Goal Attainment Scale | Baseline and approximately 2 weeks after treatment (approximately 14 weeks after baseline measurement)
  The Goal Attainment Scale is a criterion-referenced, individualized outcome measure used to assess progress on goals that are important to the child and their family. The Goal Attainment Scale is reliable, valid and responsive to change. The status of goal attainment is rated on a scale of +2 to -2 (+2 is much more than expected, -2 is much less than expected)
Change in Canadian Occupational Performance Measure | Baseline and approximately 2 weeks after treatment (approximately 14 weeks after baseline measurement)
  The Canadian Occupational Performance Measure is a valid, reliable, and sensitive assessment tool that measures the caregiver/patient's perception of the participant's performance and satisfaction on goals that are important to the child and his/her caregiver. The performance and satisfaction are rated on a scale from 1-10 (1 is low performance/satisfaction, 10 is high performance/satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Harpster, PhD, OTR/L, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available to other researchers.